CLINICAL TRIAL: NCT00541489
Title: A 13-Week, Phase 3, Multicenter, Randomized, Parallel-Group, Double-Blind, Placebo Bid and Naproxen 500 mg Bid, Controlled Study on the Efficacy on Signs and Symptoms, and Safety of Naproxcinod (HCT3012) 750 mg Bid, in Patients With Osteoarthritis of the Hip
Brief Title: Efficacy and Safety Study of Naproxcinod in Subjects With Osteoarthritis of the Hip
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NicOx (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCT3012-X-303
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Osteoarthritis; Osteoarthritis, Hip
Keywords: Osteoarthritis; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip | interventions — naproxen-n-butyl nitrate; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator): Naproxen 500 mg
  Interventions: Drug: Naproxen
- 3 (Experimental): Naproxcinod 750 mg
  Interventions: Drug: Naproxcinod

INTERVENTIONS:
Drug: Naproxcinod — 750 mg, bid
  Arms: 3
Drug: Naproxen — 500 mg, bid
  Arms: 2
Drug: Placebo — bid
  Arms: 1

SUMMARY:
To study the efficacy and safety of Naproxcinod vs. Placebo and Naproxen in the treatment of signs and symptoms of Osteoarthritis.

DETAILED DESCRIPTION:
This is a 13 week randomized, double-blind, parallel group, multicenter study comparing efficacy and safety of Naproxcinod, Placebo and Naproxen.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (40 or older) with a diagnosis of primary OA of the hip
* Must be a current chronic user of NSAIDS or acetaminophen
* Must discontinue all analgesic therapy at Screening

Exclusion Criteria:

* Uncontrolled Hypertension or Diabetes
* Hepatic or renal impairment
* Current or expected use of anticoagulant
* Clinically relevant abnormal ECG
* A history of alcohol or drug abuse
* Diagnosis of gastric or duodenal ulceration and/or history of significant gastro-duodenal bleeding, within the last 6 months
* Current medical disease, including arthritic, that could confound or interfere with the evaluation of efficacy
* Candidates for imminent joint replacement
* Participation within 30 days prior to screening in another investigational study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to show that Naproxcinod is superior to placebo in relieving OA signs and symptoms in subjects with OA of the hip

CONTACTS AND LOCATIONS:
Locations (48):
- United States (36):
  - Mobile, Alabama
  - Montgomery, Alabama
  - Tuscaloosa, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Fair Oaks, California
  - San Diego, California
  - Santa Barbara, California
  - Northglenn, Colorado
  - Coral Gables, Florida
  - Daytona Beach, Florida
  - DeLand, Florida
  - Fort Meyers, Florida
  - Jupiter, Florida
  - Louisville, Kentucky
  - Peabody, Massachusetts
  - Kalamazoo, Michigan
  - Saginaw, Michigan
  - Berlin, New Jersey
  - Dover, New Jersey
  - Rochester, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Franklin, Ohio
  - Bethany, Oklahoma
  - Duncansville, Pennsylvania
  - Penndel, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Columbia, South Carolina
  - Kingsport, Tennessee
  - Austin, Texas
  - Nederland, Texas
  - San Antonio, Texas
  - Newport News, Virginia
- Canada (12):
  - Burnaby, British Columbia
  - Coquitlam, British Columbia
  - Vancouver, British Columbia
  - Corunna, Ontario
  - Kitchener, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Québec, Quebec
  - Trois-Rivières, Quebec
  - Regina, Saskatchewan
  - Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Baerwald C, Verdecchia P, Duquesroix B, Frayssinet H, Ferreira T. Efficacy, safety, and effects on blood pressure of naproxcinod 750 mg twice daily compared with placebo and naproxen 500 mg twice daily in patients with osteoarthritis of the hip: a randomized, double-blind, parallel-group, multicenter study. Arthritis Rheum. 2010 Dec;62(12):3635-44. doi: 10.1002/art.27694. PMID 20722026
- See also: Click here to learn more about this study - Efficacy and Safety Study of Naproxcinod in Subjects with Osteoarthritis of the Hip — http://www.nicox.com